CLINICAL TRIAL: NCT03781518
Title: Mandibular Ridge Splitting With Complete Separation of the Buccal Cortical Plate Versus Khoury Shell Technique for Horizontal Augmentation of Atrophic Posterior Mandible
Brief Title: Mandibular Ridge Splitting Versus Khoury Shell Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia El- Atawy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 290316
Record Dates: First submitted 2018-11-01; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Horizontal Augmentation of Atrophic Posterior Mandible
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ridge splitting (Experimental): Mandibular ridge splitting with complete separation of the buccal cortical plate for horizontal augmentation of atrophic mandible and splinting with screws
  Interventions: Procedure: ridge splitting in group and khoury shell technique in the other group
- khoury shell technique (Active Comparator): bone block is taken from the ramus to augment deficient posterior mandible and splinting with screws
  Interventions: Procedure: ridge splitting in group and khoury shell technique in the other group

INTERVENTIONS:
Procedure: ridge splitting in group and khoury shell technique in the other group — Mandibular ridge splitting with complete separation of the buccal cortical plate for horizontal augmentation of atrophic posterior mandible in one group and the other group will receive khoury shell technique by taking bone block from the ramus

SUMMARY:
Mandibular ridge splitting with complete separation of the buccal cortical plate versus Khoury shell technique for horizontal augmentation of atrophic posterior mandible

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic mandible with residual bone width 3 to 4 mm.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* • Any pathology in the posterior mandible.

  * Heavy smokers more than 20 cigarettes per day.
  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems
  * Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Amount of horizontal bone gain (bone width) | 4 months
  measurement using CBCT

SECONDARY OUTCOMES:
Soft tissue healing | 1 months
  Dehiscence or no dehiscence

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes